CLINICAL TRIAL: NCT00529295
Title: Titrated Oral Compared With Vaginal Misoprostol for Labor Induction at Term
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: DMR95-IRB-116
Record Dates: First submitted 2007-09-13; First posted 2007-09-14 (Estimated); Last update posted 2007-09-14 (Estimated); Status verified 2006-09

CONDITIONS: Labor Induction
Keywords: misoprostol; labor induction
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Titrated oral misoprostol
  Interventions: Drug: misoprostol
- 2 (Active Comparator): Vaginal misoprostol
  Interventions: Drug: misoprostol

INTERVENTIONS:
Drug: misoprostol — Titrated oral misoprostol: one tablet of 200 microgram was dissolved in water 200 ml, and 20 ml P.O. per one hour for 4 doses, then titrated against uterine response; Vaginal misoprostol: 25 microgram per vagina

SUMMARY:
The purpose of this study was to estimate the safety and efficacy of titrated oral misoprostol compared with vaginal route for labor induction at term.

DETAILED DESCRIPTION:
Oral misoprostol absorption is more rapid and possible more predictable, with a peak serum concentration following oral administration of 34 minutes and a half-life of 20-40 minutes. Peak serum concentration for vaginal administration is 60-80 minutes, this level being sustained for up to four hours. Although the direct local effect of vaginal administration on cervical ripening may be advantageous, the shorter half-life of oral delivery may be beneficial in the event of uterine hyperstimulation.In order to avoid uterine hyperstimulation, it appears reasonable to suggest that oral misoprostol should be administered in small, frequent doses, titrated against the uterine response.

ELIGIBILITY:
Inclusion Criteria:

* 34 to 42 weeks of gestation
* live singleton
* Bishop score < or = 6
* reassuring fetal heart beat pattern

Exclusion Criteria:

* nonreassuring fetal heart beat pattern
* parity ovr five
* any contraindication to labor and/or vaginal delivery
* uterine scar
* suspected placental abruption with abnormal FHR pattern
* vaginal bleeding other than "bloody show"
* cervical dilatation of > or = 4 cm
* uterine contractions > or = 3 in 10 minutes
* significant maternal cardiac, renal or hepatic disease
* hypersensitivity to misoprostol or prostaglandin analogs

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Actual)
Dates: Start 2005-06; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
The interval from the first misoprostol dose to vaginal delivery and the percentage of women who delivered infants vaginally within 12 and 24 hours of induction. The incidence of tachysystole, hypertonus, uterine hyperstimulation and neonatal outcomes. | within the first week after delivery

SECONDARY OUTCOMES:
Total dosage of misoprostol and the rate of women given oxytocin, cesarean section and induction failure. | The days during induction

CONTACTS AND LOCATIONS:
Overall Officials: Shi-Yann Cheng, M.D., Principal Investigator — Chinal Medical University Beigang Hospital
Locations (1):
- China Medical University Beigang Hospital, Douliu, Taiwan

REFERENCES:
- [Result] Hofmeyr GJ, Alfirevic Z, Matonhodze B, Brocklehurst P, Campbell E, Nikodem VC. Titrated oral misoprostol solution for induction of labour: a multi-centre, randomised trial. BJOG. 2001 Sep;108(9):952-9. doi: 10.1111/j.1471-0528.2001.00231.x. PMID 11563466
- [Derived] Kerr RS, Kumar N, Williams MJ, Cuthbert A, Aflaifel N, Haas DM, Weeks AD. Low-dose oral misoprostol for induction of labour. Cochrane Database Syst Rev. 2021 Jun 22;6(6):CD014484. doi: 10.1002/14651858.CD014484. PMID 34155622
- [Derived] Cheng SY, Ming H, Lee JC. Titrated oral compared with vaginal misoprostol for labor induction: a randomized controlled trial. Obstet Gynecol. 2008 Jan;111(1):119-25. doi: 10.1097/01.AOG.0000297313.68644.71. PMID 18165400